CLINICAL TRIAL: NCT01329055
Title: International Comparison of Evolution of Clinical and Laboratory Parameters in Chronic Hemodialysis Patients
Brief Title: Events Before Death
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Collaborators: Fresenius Medical Care North America (Industry); Maastricht University (Other); University of California (Other); Medical University Innsbruck (Other)
Responsible Party: Peter Kotanko MD, Renal Research Institute
Other Study IDs: 10-119
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis patients

SUMMARY:
Previous studies of the patients treated in RRI clinics suggest that hemodialysis patients undergo a certain consistent predictable pattern at the initiation of dialysis and before death. This pattern can be described as a group of patterns of patients' biological markers over a few months after starting dialysis and several months prior to death. Additional patterns can be observed that occur with changes in seasons or time of day. The aim of this study is to compare these patterns in patients treated in FMC-Asia, FMC-Europe, FMC-South America, and RRI-US populations. Noting that patterns in patient parameters are similar across continents, climates, and geographic variations only further accentuates the importance in the models that can predict patients' survival and provide an opportunity for timely intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis vintage 2+ months

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2000-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Date of death | 10 years and 5 months
  The main purpose of the study is developing an alert system that will help dialysis providers recognize patients who are at increased risk of death (or hospitalization). This alert system will be developed and can be utilized in patients treated all over the world.

SECONDARY OUTCOMES:
Hospitalizations | January 2000 - May 2010

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Institute, New York, New York, United States